CLINICAL TRIAL: NCT02416063
Title: Caudal Versus Intravenous Dexmedetomidine for Caudal Analgesia in Children: A Randomised Controlled Double Blind Study
Brief Title: Caudal Versus Intravenous Dexmedetomidine for Caudal Analgesia in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Khaled Radian Al-zaben, Dr, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Faculty of medicine-JU
Record Dates: First submitted 2015-03-12; First posted 2015-04-14 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- caudal Dexmedetomidine (Active Comparator): Drug:Caudal Bupivacaine 0.25% 1ml/kg .
  Drug:caudal Dexmedetomidine 1μg /kg.
  Intravenous :10 ml normal saline
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Caudal Dexmedetomidine
- Intravenous Dexmedetomidine (Active Comparator): Drug:Caudal bupivacaine 0.25% 1ml/kg
  Drug: Intravenous dexmedetomidine 1µg/kg in a 10 ml volume normal saline
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Intravenous dexmedetomidine
- Placebo (Placebo Comparator): Caudal: bupivacaine 0.25% 1ml/kg .
  Intravenous: 10 ml Normal saline
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Caudal Dexmedetomidine — Drug:Caudal bupivacaine 0.25% 1ml/kg
  Drug: Caudal dexmedetomidine 1µg/kg
  Intravenous: 10 ml normal saline
  sevoflurane Induction and maintenance of anesthesia
  Other Names: dexmedetomidine; Precedex
  Arms: caudal Dexmedetomidine
Drug: Intravenous dexmedetomidine — Drug:Caudal bupivacaine 0.25% 1ml/kg.
  Drug:Intravenous dexmedetomidine1 μg /kg in a total volume of 10 ml
  sevoflurane Induction and maintenance of anesthesia
  Other Names: precedex
  Arms: Intravenous Dexmedetomidine
Drug: Placebo — Drug:Caudal bupivacaine 0.25% 1ml/kg
  Intravenous: Normal saline 10 ml
  sevoflurane Induction and maintenance of anesthesia
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
The aim of this prospective randomized double-blind study was to compare the analgesic efficacy and the side effects of dexmedetomidine (1 µg.kg-1) co-administered with bupivacaine for caudal analgesia or intravenously in children undergoing infra-umbilical surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is used increasingly in pediatric anesthesia practice to prolong the duration of action of caudal block with a local anesthetic agent.But which route of administration of dexmedetomidine is the most beneficial remains unknown.

The investigators performed prospective randomized double-blind study to compare the effects of caudal dexmedetomidine with intravenous dexmedetomidine on postoperative analgesia after caudal bupivacaine in children undergoing infra-umbilical surgery.

75 children (ASAⅠorⅡ,aged 1-6 yr) undergoing infra-umbilical surgery were included in this study. Anesthesia was induced with sevoflurane via a facemask, followed by placement of a laryngeal mask airway. Anesthesia was maintained with sevoflurane 2-3% in oxygen-air.Then,caudal block was applied. Patients were randomly assigned in three groups. Group B-Dcau (n = 25): Caudal bupivacaine 0.25% 1ml/kg plus dexmedetomidine 1µg/kg and 10 ml normal saline i.v.;Group B-Div (n = 25): bupivacaine 0.25% 1ml/kg and dexmedetomidine 1µg/kg(10 ml)i.v.;Group B(n = 25): bupivacaine 0.25% and 10 ml normal saline intravenous

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) - I
* Scheduled for lower abdominal and perineal surgery
* Under general anesthesia

Exclusion Criteria:

* Hypersensitivity to any local anesthetics
* Patient has history of allergy, intolerance, or reaction to dexmedetomidine
* Infections at puncture sites
* Bleeding diathesis
* Preexisting neurological disease
* Children with uncorrected cardiac lesions
* Children with heart block

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time to first analgesic requirement | 24 hours
  Time to first rescue medication. The time from end of surgery to the first requirement of postoperative analgesia,pain score ≥4

SECONDARY OUTCOMES:
Postoperative behaviour scores | 2 hours
  behaviour score was recorded throughout the post-anesthesia care unit stay at 15-minute time intervals.
Sevoflurane concentration | 1 hour
  Sevoflurane concentration required to maintain Bispectral Index (BIS) monitor reading between 40 and 60
Blood pressure Perioperative blood pressure readings | 2 hours
  Perioperative blood pressure readings
Heart Rate | 2 hours
  Perioperative heart rate readings
the incidence of emergence agitation | 2 hours
  Participants will be followed for the duration of PACU stay, an expected average of 2 hours
Postoperative pain scores | 24 hours
  postoperative pain score will be assessed over 24 hours
Side effects | 24 hours
  side effects including nausea, vomiting and urinary retention and lower limb weakness

CONTACTS AND LOCATIONS:
Overall Officials: khaled R Al-zaben, Principal Investigator — University of Jordan

REFERENCES:
- [Background] Zhang C, Hu J, Liu X, Yan J. Effects of intravenous dexmedetomidine on emergence agitation in children under sevoflurane anesthesia: a meta-analysis of randomized controlled trials. PLoS One. 2014 Jun 16;9(6):e99718. doi: 10.1371/journal.pone.0099718. eCollection 2014. PMID 24932765
- [Background] Guler G, Akin A, Tosun Z, Ors S, Esmaoglu A, Boyaci A. Single-dose dexmedetomidine reduces agitation and provides smooth extubation after pediatric adenotonsillectomy. Paediatr Anaesth. 2005 Sep;15(9):762-6. doi: 10.1111/j.1460-9592.2004.01541.x. PMID 16101707
- [Background] Al-Zaben KR, Qudaisat IY, Al-Ghanem SM, Massad IM, Al-Mustafa MM, Al-Oweidi AS, Abu-Halaweh SA, Abu-Ali HM, Saleem MM. Intraoperative administration of dexmedetomidine reduces the analgesic requirements for children undergoing hypospadius surgery. Eur J Anaesthesiol. 2010 Mar;27(3):247-52. doi: 10.1097/EJA.0b013e32833522bf. PMID 19952754
- [Background] Kim NY, Kim SY, Yoon HJ, Kil HK. Effect of dexmedetomidine on sevoflurane requirements and emergence agitation in children undergoing ambulatory surgery. Yonsei Med J. 2014 Jan;55(1):209-15. doi: 10.3349/ymj.2014.55.1.209. PMID 24339309
- [Background] She YJ, Xie GT, Tan YH, Kuang XH, Yu GF, Lian GH, Song XR. A prospective study comparing the onset and analgesic efficacy of different concentrations of levobupivacaine with/without dexmedetomidine in young children undergoing caudal blockade. J Clin Anesth. 2015 Feb;27(1):17-22. doi: 10.1016/j.jclinane.2014.09.005. Epub 2014 Nov 21. PMID 25468576
- [Background] Schnabel A, Reichl SU, Poepping DM, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of intraoperative dexmedetomidine for acute postoperative pain in children: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2013 Feb;23(2):170-9. doi: 10.1111/pan.12030. Epub 2012 Oct 9. PMID 23043461
- [Background] Fares KM, Othman AH, Alieldin NH. Efficacy and safety of dexmedetomidine added to caudal bupivacaine in pediatric major abdominal cancer surgery. Pain Physician. 2014 Sep-Oct;17(5):393-400. PMID 25247897